CLINICAL TRIAL: NCT05086874
Title: A Real-world Retrospective Study on the Effectiveness and Safety of Butylphthalide in the Treatment of Ischemic Stroke
Brief Title: Using Real-world Evidence to Analyze the Clinical Effects and Adverse Events of Butylphthalide in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Xin Huang (Other)
Responsible Party: Sponsor-Investigator, Xin Huang, Chief Pharmacist, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: QFS-HX-2021-DBT-HGX-001
Record Dates: First submitted 2021-09-25; First posted 2021-10-21 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Cerebral Infarction; Brain Infarction; Brain Ischemia; Nervous System Diseases; Central Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases
Keywords: butylphthalide; Ischemic Strokes; Real world research
MeSH Terms: conditions — Stroke; Cerebral Infarction; Brain Infarction; Brain Ischemia; Nervous System Diseases; Central Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Ischemic Stroke | interventions — 3-n-butylphthalide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: A group of patients with ischemic stroke, treated with butylphthalide
  Interventions: Other: butylphthalide
- Non-exposed group: A group of patients with ischemic stroke, treated with Edaravone

INTERVENTIONS:
Other: butylphthalide — Observational only and no predesigned interventions in this study
  Other Names: observational only ,no intervention
  Groups: Exposed group

SUMMARY:
This is a retrospective, multi-center, real-world study. The researchers plan to include 10,000 cases of ischemic stroke patients using butylphthalide and 10,000 cases of ischemic stroke patients using Edaravone. The main purpose is to analyze the effectiveness and safety of butylphthalide and establish the drug risk assessment management plan.

DETAILED DESCRIPTION:
Ischemic stroke is a type of syndrome in which blood supply to the brain is impaired due to various reasons, leading to local brain tissue ischemia, hypoxic necrosis, and corresponding neurological deficits. It has a high incidence, high morbidity and disability. Features of high recurrence rate.

Butylphthalide can improve the damage of central nervous system in patients with acute ischemic stroke, and can promote the improvement of patients with neurological deficits. Regarding butylphthalide in the treatment of ischemic stroke, there is still a lack of big data research based on the efficacy and safety of the real world.

Therefore, it is planned to include 10,000 patients who used butylphthalide or Edaravone in five hospitals from 2019 to 2021, and record the basic information of the patients, medication status and related test results. The data was cleaned, sorted and analyzed to evaluate the effectiveness and safety of butylphthalide in the treatment of ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* From January 2019 to August 2021, clinicians diagnosed patients with ischemic stroke requiring hospitalization.

Exclusion Criteria:

* Patients who are unable to obtain information such as medical advice, laboratory test results, etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Doctors diagnosed with ischemic stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 81292 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events | 90days
  The probability of unanticipated and adverse medical events after the patient receives medication, but it does not necessarily have a causal relationship with the treatment

SECONDARY OUTCOMES:
NIHSS | 90days
  NIH stroke scale (NIHSS) to assess the degree of neurological deficit in stroke patients. The score ranges from 0 to 42 points, the higher the score, the more severe the nerve damage. Patients with a baseline assessment of> 16 points are likely to die, while those with a score of <6 are likely to recover well; for each additional point, the probability of a good prognosis is reduced by 17%
mRS | 90days
  Modified Rankin scale (mRS) is an indicator of the efficacy of functional disability. The score ranges from 0 to 5 points, and the clinical score will be increased to 6 points to indicate death. The higher the score, the more disability the patient is.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Huang, Study Director — Qianfoshan Hospital
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Jinan, Shandong Provincial, China

IPD SHARING:
Plan to Share IPD: Undecided
Haven't decided yet